CLINICAL TRIAL: NCT05501405
Title: Brain and Oculometric Markers of Emotional Facial Expression Recognition Deficits Associated With Autistic and Psychotic Symptoms
Brief Title: Brain and Oculometric Markers of Emotional Facial Expression Recognition Deficits
Acronym: FERmarkers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator départure
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-A01367-34
Record Dates: First submitted 2022-03-21; First posted 2022-08-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Autism; Psychotic Disorders
MeSH Terms: conditions — Autistic Disorder; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Brain and eyetracking markers of deficits in recognition of emotional facial expression and associated autistic and/or psychotic disorders
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Schizophrenic patients (Experimental): Electroencephalogram and eye-tracking recordings Behavorial tests
  Interventions: Other: Electroencephalogram and eye-tracking recordings
- Autism Spectrum Disorder (ASD) patients (Experimental): Electroencephalogram and eye-tracking recordings
  Interventions: Other: Electroencephalogram and eye-tracking recordings
- 22q11.2 DS patients (Experimental): Electroencephalogram and eye-tracking recordings Behavorial tests
  Interventions: Other: Electroencephalogram and eye-tracking recordings
- Williams syndrome patients (Experimental): Electroencephalogram and eye-tracking recordings Behavorial tests
  Interventions: Other: Electroencephalogram and eye-tracking recordings
- Präder Willi syndrome patients (Experimental): Electroencephalogram and eye-tracking recordings Behavorial tests
  Interventions: Other: Electroencephalogram and eye-tracking recordings
- Control participants (Active Comparator): Electroencephalogram and eye-tracking recordings Behavorial tests
  Interventions: Other: Electroencephalogram and eye-tracking recordings

INTERVENTIONS:
Other: Electroencephalogram and eye-tracking recordings — Participants will perform two tasks: recognize the expression (explicit recognition of the expression) or detect the change in color of the cross (implicit processing of the expression). Each participant will perform two tasks x 6 models x 5 expressions, i.e. 60 stimulations, for a stimulation duration of approximately 30 minutes.
  Recognition of the emotional facial expression with a choice among 5 possibilities. Two neutral faces of the same person will be presented side by side. When the participant has looked at the central fixation cross for one second, one of the two faces will produce an expression. The participant will have to indicate as quickly as possible which expression it is, while his or her eye movements are recorded. Each participant will have to recognize 5 expressions x 8 models, i.e. 40 trials for a duration of approximately 5 to 10 minutes
  Other Names: Behavorial tests

SUMMARY:
Disorders in the recognition of emotional facial expressions are part of the social cognition disorders described in several diseases. They are notably present in a quasi-systematic way in diseases associated with socio-emotional behavior disorders, such as schizophrenia and autism. They are also found in some genetic syndromes with atypical neurodevelopment. In previous studies, the investigators adopted the FPVS-EEG approach to investigate facial emotion discrimination abilities in typical and atypical developing populations. the investigatorshave shown that, in typical adults, the neural response to facial expressions emerges as emotional intensity parametrically increases. A time-domain analysis revealed three components, with the first two increasing linearly with expressive intensity, and the third (beyond 300 ms) showing categorical sensitivity to increasing expressive intensity. The investigators have already successfully extended this approach to the investigation of patients, such as those with 22q11.2 syndrome. The brain response to facial expression was reduced by approximately 36% in these patients, revealing impaired visual coding of emotional facial signals. In this study, response amplitude was associated with positive symptom severity, indicating a potential endophenotype for psychosis risk. Here, the investigators study the implementation of high-level processes and the top-down effect it should have on the response of occipitotemporal regions to identify altered brain markers in schizophrenic patients, but also in other populations with expression recognition deficits (autistic, 22q11.2, in particular). The implementation of compensatory strategies that should result in an increased exploration of the lower part of the face at the oculometric level will also be studied.

DETAILED DESCRIPTION:
Disorders in the recognition of emotional facial expressions are part of the social cognition disorders described in several pathologies. In particular, they are almost systematically present in pathologies associated with socio-emotional behavior disorders, such as schizophrenia and autism. They are also found in certain genetic pathologies with atypical neurodevelopment .

Recently, it has been suggested to use a new approach to better understand the brain specificity of populations with face recognition difficulties: the Fast Periodic Visual Stimulation (FPVS) approach coupled with electroencephalography (FPVS-EEG) . This has been done successfully for Autism Spectrum Disorder. The investigators have also done this for 22q11.2 syndrome . This approach has proven to be particularly well suited to the study of atypical populations. However, studies to date have investigated the implicit processing of emotional facial expression. The role of top-down mechanisms related to the task remains to be studied.

Moreover, in these different diseases, difficulties in facial emotion recognition are furthermore associated with abnormalities in the visual exploration of facial features. Some profiles (looking at the lower part) might reflect compensatory strategies to compensate for difficulties in perceiving the whole face or the upper part (i.e., the eye region). Other patterns (disorganized exploration) could reflect the prevalence of psychotic signs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a genetic condition with psychiatric expression (22q11.2 microdeletion syndrome, Williams syndrome, Präder-Willi syndrome)
* Individuals with schizophrenia according to DSM-5 criteria
* Individuals with Autism Spectrum Disorder (ASD) according to DSM-5 criteria
* Individuals between the ages of 10 and 50
* French native language
* Psychotropic treatment unchanged during the month preceding inclusion
* Stable symptomatology
* Individuals having given their informed consent to participate in the study (consent of legal tutors for minors or under tutorship

Exclusion Criteria:

* Recent addiction, excluding tobacco addiction (according to DSM-5 criteria)
* Neurological disorders of vascular, infectious or neurodegenerative origin for patients with schizophrenia or ASD
* Uncorrected visual acuity disorder
* Use of somatic medications that have a cerebral or psychological impact (e.g. corticosteroids)
* Pregnant women

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Fast Periodic Visual Stimulation Task (FPVS-EEG) | 48 months
  Fast periodic visual stimulation (FPVS) allows the recording of objective brain responses of human face categorization (i.e., generalizable face-selective responses) with high signal-to-noise ratio.The electrical activity of the brain will be collected using an electroencephalography system (EEG; systems used: ANT and BioSemi) to study the cerebral frequency response to the regular occurrence of facial expressions.

SECONDARY OUTCOMES:
Eye-tracking task | 48 months
  Ocular exploration in the recognition of emotional facial expressions Use of the Eye-tracker (Tobii brand, 250 Hz frequency) to record the participants' eye activity. The task will consist of presenting the neutral face of a person on either side of a fixation cross. The participant will have to stare at the fixation cross for one second to trigger the replacement of one of the two neutral faces by the face of the same person expressing an emotion and will have to identify, as quickly as possible, which of the 5 emotions (anger, disgust, fear, happiness or sadness) is expressed by the face. After the calibration of the participant's gaze, the latter will carry out a training session of 10 trials [2 models (1 woman/1 man) x 5 expressions per model], then an experimental session of 40 trials (6 models (3 women/3 men) x 5 expressions) organized in 2 blocks of 20 trials. The presentation of the trials will be done in a random order.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCK NICOLAS, PhD, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- centre de réhabilitation - Hôpital le Vinatier, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No